CLINICAL TRIAL: NCT06353100
Title: Chronic Pain in the General Population of Chile: Longitudinal Study
Brief Title: Chronic Pain in the General Population of Chile
Acronym: RDC
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Chilean Safety Association (ACHS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 230602006
Record Dates: First submitted 2024-02-05; First posted 2024-04-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain; Migraine Disability; Neuropathic Pain; Fibromyalgia; Depression, Anxiety; Self Harm; Insomnia; Loneliness
Keywords: Chronic pain; Depression; Anxiety; Incidence; Prevalence
MeSH Terms: conditions — Chronic Pain; Neuralgia; Fibromyalgia; Depression; Anxiety Disorders; Self-Injurious Behavior; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Longitudinal analysis group 1 (no pain): Participants (general population residing in urban areas of Chile aged 18 years or more) not reporting chronic pain in march 2023 or march 2024
- Longitudinal analysis group 2 (incident chronic pain): Participants (general population residing in urban areas of Chile aged 18 years or more) not reporting chronic pain in march 2023 but reporting chronic pain in march 2024
- Longitudinal analysis group 3 (remitted chronic pain): Participants (general population residing in urban areas of Chile aged 18 years or more) reporting chronic pain in march 2023 but not reporting it in march 2024
- Longitudinal analysis group 4 (chronic pain at follow up): Participants (general population residing in urban areas of Chile aged 18 years or more) reporting chronic pain in march 2023 and march 2024

SUMMARY:
The present study seeks to follow up the cohort of adults representative of Chile's urban population whose levels of chronic pain were evaluated in March 2023 (baseline) as part of the Mental Health Thermometer (MHT) study. The study consists of a 12 month follow-up telephone interview to assess parameters of chronic pain (CP) and subtypes, mental and physical health, lifestyle and adversity and work characteristics.

The study objectives are as follows:

1. Estimate the prevalence of CP and subtypes in the general population
2. Explore the association between mental health indicators, perceived work stress and presence of CP in the population.
3. Investigate the impact of CP (functional, occupational and social) among the subset of participants reporting CP
4. Describe the use of management strategies in those who suffer from CP.

DETAILED DESCRIPTION:
I. Aims of the study:

1. Estimate the prevalence of chronic pain (CP) and subtypes in the
2. Explore the association between mental health indicators, perceived work stress and the presence of CP in the urban population of Chile.
3. Asses the functional, occupational and social impact of CP in Chile´s urban population reporting CP.
4. Describe the use of management strategies in those who suffer from CP.

II. Design:

The design is longitudinal prospective and involves following up the same group of participants from the MHT study to monitor their mental health and CP parameters.

III. Study variables include:

3.1. Main outcome measures (instrument): Presence of chronic pain in the last 3 months, Severity of chronic pain (Chronic pain grade questionnaire; CPG), chronic pain interference in daily activities, social activities and work (CPG), depression (Patient Health Questionnaire; PHQ-9), anxiety (General Anxiety Disorder (GAD-7) 3.2. Secondary outcome measures: chronic pain management strategies, migraine disability (Migraine Disability Assessment, MIDAS), neuropathic pain (Neuropathic pain DN4 Questionnaire; DN4), fibromyalgia (Fibromyalgia Survey Questionnaire; FSQ), insomnia (Insomnia Severity Index; ISI), loneliness (3-item UCLA Loneliness Scale; R-UCLA) 3.3. Variables of interest: job-relates stress (Copenhagen Burnout Inventory; CBI), childhood adversity (Adverse childhood experiences; ACE), negative life events.

IV. Groups:

For the longitudinal analysis, participants will be classified into four groups:

* Group 1 (no pain): participants who do not declare CP at baseline or follow-up
* Group 2 (incident): participants who do not declare CP at baseline but declare it at follow-up.
* Group 3 (remitted): participants who declare CP at baseline but do not declare it at follow-up.
* Group 4 (chronic pain at follow-up): participants who declare CP at baseline and follow-up

V. Analysis plan:

5.1. Cross-sectional analysis (at follow-up)

* Prevalence of CP will be calculated (with 95% confidence interval (CI)) for the Chilean urban population by sex, age group and employment status (aim 1).
* Prevalences of the most common CP syndromes (i.e. migraine, fibromyalgia, neuropathic pain) with 96% CI will also be calculated.
* In the subset of the population with CP, descriptive analyzes will be carried out (percentages, means and standard deviation) of the interference levels (aim 3) and chronic pain management strategies (aim 4) by sex, age group and employment status.
* Calculation of Odds Ratios (ORs) with 95% CI for the main mental health variables associated with the presence of CI (i.e. symptoms of depression and anxiety) and for work variables (i.e. work-related stress), using logistic regression, adjusting for age, sex, physical health characteristics (aim 2).

5.2. Longitudinal analysis (baseline and follow-up)

* The database will be integrated with the baseline data and based on the distribution of certain sociodemographic and health variables in the two times, an attrition analysis will be carried out to conclude on the selective loss of subjects.
* Four groups will be created according to the pain trajectory between the two measurement points (see group section) and the proportion of new cases in the 12 months will be calculated (i.e. annual incidence).
* The difference in the chronic pain intensity reported at the measurement points will be calculated.
* Several multilevel models will be analyzed to examine the relationship between mental health (PHQ-9 and GAD- 7), sleep difficulties (ISI), perception of loneliness (UCLA-R), health variables (alcohol consumption, tobacco, body mass) and work variables (i.e. job satisfaction, work-related stress) and changes in the magnitude of perceived CP at 12 months, using linear and non-linear mixed effects models (aim 3).

ELIGIBILITY:
Inclusion Criteria:

* General population
* Residence in urban areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community survey in Chile
Sampling Method: Probability Sample
Enrollment: 2365 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Chronic pain (past 3 months) | Baseline and 12-month follow-up
  Participants will be asked "Have you had constant or frequent pain [most of the day] during the past 3 months?" and asked to identify the average and maximum intensity of pain in that period using a visual analogue scale (VAS) from 0 to 10. Only participants with an average pain of 4 or more will be classified as having significant chronic pain.
Depression (2 weeks) | Baseline and 12-month follow-up
  As measured by the Patient Health Questionnaire (PHQ-9). Total scores on the PHQ-9 range from 0 to 27 and higher scores indicate higher symptoms of depression.
Anxiety (2 weeks) | Baseline and 12-month follow-up
  As measured by the General Anxiety Disorder (GAD-7). Total scores on the GAD-7 range from 0 to 21 and higher scores indicate higher symptoms of anxiety.

SECONDARY OUTCOMES:
Migraine Disability | 12-month follow-up
  As measured by the MIDAS (Migraine Disability Assessment). Total scores on the MIDAS range from 0 to 20 and higher scores indicate higher disability.
Neuropathic Pain | Baseline and 12-month follow-up
  As measured by the DN4 (Neuropathic pain DN4 Questionnaire). Total scores on the DN4 range from 0 to 10 and Scores ≥ 4/10 indicate neuropathic pain.
Fibromyalgia | 12-month follow-up
  As measured by the Fibromyalgia Survey Questionnaire (FSQ). The possible score ranges from 0 to 31 points. A score equal to or greater than 13 points is consistent with a diagnosis of fibromyalgia.
Self harm (2 weeks) | Baseline and 12-month follow-up
  As measured by item 9 (Thoughts that you would be better off dead or of hurting yourself in some way) of the Patient Health Questionnaire (PHQ-9).
Insomnia (2 weeks) | Baseline and 12-month follow-up
  As measured by the Insomnia Severity Index (ISI). Responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia.
Loneliness | Baseline and 12-month follow-up
  As measured by the 3-item University of California, Los Angeles Loneliness Scale (R-UCLA). Total scores range from 3 to 9 and higher scores indicate higher perceived loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Errazuriz, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Yes
The anonymized database and codebook will be made available to researcher in the Dataverse website
Supporting Information: Study Protocol, ICF
Time Frame: Upon first manuscript submission
Access Criteria: For researchers